CLINICAL TRIAL: NCT01170065
Title: A Phase II Open Label, Roll Over Study of the Long Term Tolerability, Safety and Efficacy of Oral BIBF 1120 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Roll Over Study From 1199.30 BIBF 1120 in Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.35; 2009-013788-21 (EudraCT Number)
Record Dates: First submitted 2010-07-06; First posted 2010-07-27 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — nintedanib

ARMS (4):
- BIBF 1120 low qd (Experimental): Low dose BIBF 1120 once daily
  Interventions: Drug: BIBF 1120
- BIBF 1120 low bid (Experimental): Low dose BIBF 1120 twice daily
  Interventions: Drug: BIBF 1120
- BIBF 1120 medium bid (Experimental): Intermediate dose BIBF 1120 twice daily
  Interventions: Drug: BIBF 1120
- BIBF 1120 high bid (Experimental): High dose BIBF 1120 twice daily
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120 — Intermediate dose BIBF 1120 twice daily
  Arms: BIBF 1120 medium bid
Drug: BIBF 1120 — High dose BIBF 1120 twice daily
  Arms: BIBF 1120 high bid
Drug: BIBF 1120 — Low dose BIBF 1120 twice daily
  Arms: BIBF 1120 low bid
Drug: BIBF 1120 — Low dose BIBF 1120 once daily
  Arms: BIBF 1120 low qd

SUMMARY:
The aim of this trial is to offer continuation of BIBF 1120 treatment for patients with Idiopathic Pulmonary Fibrosis (IPF) who have completed a prior clinical trial with that drug.

The primary objective will be to establish the long term tolerability and safety profile of BIBF 1120 in Idiopathic Pulmonary Fibrosis (IPF).

As a secondary objective the effects of long term treatment with BIBF 1120 on survival as well as safety and efficacy parameters will be investigated in an open-label, not randomized, un-controlled design.

ELIGIBILITY:
Inclusion criteria:

1. Patient with a primary diagnosis of IPF (according to the 2000 American Thoracic Society/European Respiratory Society (ATS/ERS) criteria, who are willing to continue trial medication.
2. Written informed consent signed prior to entry into the study, in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local law
3. Completion of 1199.30 study and still under treatment (i.e. not discontinued in parent trial)

Exclusion criteria:

1. Any disease that may put the patient at risk when participating in this trial. Reconsider carefully all exclusion criteria of trial 1199.30. However, patients may qualify for participation even though exclusion criteria may have been met during the course of participation in 1199.30, if the investigator's benefit-risk assessment remains favourable.
2. Participation in another experimental clinical trial (except 1199.30) in the last 8 weeks.
3. Women who are breast feeding or of child bearing potential not using a highly effective method of birth control for at least one month prior to inclusion and at least 10 weeks after end of active therapy.

   Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1 % per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some Intra Uterine Devices (IUDs), sexual abstinence or vasectomized partner. Female patients will be considered of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
4. Sexually active males not committing to using condoms during the course of the study and at least 10 weeks after the end of active therapy (except if their partner is not of childbearing potential).
5. Patients who require full-dose anticoagulation (e.g. vitamin K antagonists, heparin, hirudin etc).
6. Patients who require full-dose antiplatelet (e.g. acetyl salicylic acid, clopidogrel etc) therapy.
7. Known or suspected active alcohol or drug abuse.
8. Patient not compliant in previous trial, with trial medication or trial visits.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2010-06-25 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (57):
- INSARES, Mendoza, Argentina
- Australia (3):
  - Respiratory Clinical Trial Pty Ltd., Glen Osmond, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Royal Perth Hospital-Lung Transplant Unit, Perth, Western Australia
- Belgium (3):
  - ULB Hopital Erasme, Brussels
  - UZ Leuven, Leuven
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir
- Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Brazil
- Special. Hospital for Active Treatment, Sv. Sofia 2nd Clinic, Sofia, Bulgaria
- Canada (2):
  - QEII Health Sciences Centre (Dalhousie University), Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
- Instituto Nacional del Tórax, Santiago, Chile
- China (4):
  - Beijing Chao-Yang Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Nanjing Drum Tower Hospital, Nanjing
  - Shanghai Pulmonary Hospital, Shanghai
- Czechia (2):
  - University Hospital Na Bulovce, Prague, Prague
  - Masaryk Hospital, Usti nad Labem, Ústí nad Labem
- France (6):
  - HOP Avicenne, Bobigny
  - HOP Dijon, Pneumo, Dijon, Dijon
  - HOP Calmette, Lille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - HOP Bichat, Paris
- Germany (6):
  - Klinik Donaustauf, Donaustauf
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Freiburg, Freiburg/Breisgau
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München - Campus Großhadern, München
- Greece (2):
  - University General Hospital of Evros, Alexandroupoli
  - University Hospital of Heraklion, University Pulmonology Cl, Heraklion
- Hungary (2):
  - Csongrad County's Hosp., Deszk
  - University of Pecs, 1st internal Med. Dept., Pulmonology, Pécs
- Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (8):
  - Ospedale C. G. Mazzoni, Ascoli Piceno
  - Osp. S. Giuseppe Fatebenefratelli, Milan
  - Università di Modena e Reggio Emilia, Modena
  - Università Federico II, Napoli
  - Pol. Universitario Tor Vergata, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - Università di Perugia, Terni
  - Ospedale di Cattinara, Trieste
- Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas, Distrito Federal, Mexico
- St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein, Netherlands
- Portugal (4):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - CHLN, EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Lisboa Norte Hospital Pulido Valente, Lisbon
  - Centro Hospitalar São João,EPE, Porto
- Russia (2):
  - Central Scientific Research Insitute of Tuberculosis, Moscow
  - Scientific Research Institute of Pulmonology, Saint Petersburg
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Dr. Peset, Valencia
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - The Medicines Evaluation Unit, Manchester
  - Southmead Hospital, Westbury on Trym

REFERENCES:
- [Derived] Richeldi L, Kreuter M, Selman M, Crestani B, Kirsten AM, Wuyts WA, Xu Z, Bernois K, Stowasser S, Quaresma M, Costabel U. Long-term treatment of patients with idiopathic pulmonary fibrosis with nintedanib: results from the TOMORROW trial and its open-label extension. Thorax. 2018 Jun;73(6):581-583. doi: 10.1136/thoraxjnl-2016-209701. Epub 2017 Oct 9. PMID 28993537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment groups are displayed according to dose at randomisation in 1199.30 (NCT00514683).
Pre-assignment Details: Patients were not randomised to study medication in trial 1199.35 but were to receive open-label nintedanib, either at the dose received in period 2 of parent trial 1199.30 (NCT00514683) or they could increase their dose to nintedanib 150 mg twice daily (bid) after implementation of protocol amendment 1.
Groups:
- Placebo: Patients were treated with oral administration of placebo in period 1 of the parent trial and with soft gelatine capsules of Nintedanib 50 mg once daily (qd) in the second period of the 1199.30 (parent trial). In the 1199.35 trial they could remain on this last dose or increase to Nintedanib 150 mg twice daily (bid)
- Nintedanib 50 mg- 100 mg: Patients were treated with oral administration of soft gelatine capsules of Nintedanib 50 mg qd, 50 mg bid or 100 mg bid in the parent trial. In the 1199.35 trial they could remain on their last dose in the parent trial or increase to Nintedanib 150 mg bid.
- Nintedanib 150 mg: Patients were treated with oral administration of soft gelatine capsules of Nintedanib 150 mg bid and could step down to 100 mg bid. In the 1199.35 trial they could remain on their last dose in the parent trial.
Period: Overall Study
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Started | 37 | 126 | 35
Completed | 9 (Planned observation time is from first trial drug intake to follow-up visit) | 34 (Planned observation time is from first trial drug intake to follow-up visit) | 9 (Planned observation time is from first trial drug intake to follow-up visit)
Not Completed | 28 | 92 | 26
Not completed — Adverse Event | 17 | 50 | 10
Not completed — Lost to Follow-up | 1 | 4 | 1
Not completed — Consent withdrawn, not due to AE | 2 | 4 | 2
Not completed — Reason other than specified | 3 | 8 | 3
Not completed — Ongoing after planned observation time | 5 | 26 | 10

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set which included all patients who received at least 1 dose of open-label study medication in trial 1199.35
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg | Total
Number analyzed (Participants) | 37 | 126 | 35 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.3) | 65.4 (8.6) | 65.2 (7.2) | 65.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 36 | 7 | 57
  Male | 23 | 90 | 28 | 141

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is the total amount of air exhaled during the lung function test.
  For this endpoint reported means represent the adjusted rate.
Time Frame: From first drug administration in 1199.35 until database lock 15Oct2015, up to 61.8 Months
Population: The full analysis set (FAS): which included all patients in the treated set who provided baseline data (for the first trial visit) for at least 1 endpoint in trial 1199.35
Measure: Mean (Standard Error); unit: milliliters per year (mL/ yr)
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
milliliters per year (mL/ yr) | -129.0 (29.47) | -137.5 (14.60) | -132.9 (28.22)

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the first intake of nintedanib in trial 1199.35 to death.
  For presentation of overall survival results, Kaplan-Meier estimates and confidence intervals (using Greenwood variance formula) for the overall on-treatment survival is calculated within each treatment arm.
Time Frame: From first drug administration in 1199.35 until database lock 15Oct2015, up to 61.8 Months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
percentage of participants | 37.4 (29.47) [16.8 to 58.0] | 46.8 (14.60) [35.3 to 58.4] | 66.2 (28.22) [46.9 to 85.5]

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the time from the first nintedanib intake in trial 1199.35 to disease progression.
  For presentation of progression-free survival results, Kaplan-Meier estimates and confidence intervals (using Greenwood variance formula) for the overall on-treatment progression-free survival is calculated within each treatment arm.
Time Frame: From first trial drug intake in 1199.35 to disease progression; up to 61.8 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
percentage of participants | 9.6 (29.47) [0.0 to 22.0] | 3.5 (14.60) [0.0 to 7.4] | 12.2 (28.22) [0.0 to 24.9]

4. Secondary Outcome: Annual Rate of Decline in Haemoglobin Corrected Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) Decrease
Description: Haemoglobin corrected DLCO decrease was a secondary endpoint for the trial. It was considered important that all investigators used the same method of testing and recording data at each visit for each patient.
  Haemoglobin corrected DLCO was calculated for each patient using the following formulae:
  Males: Hb corrected DLCO = measured DLCO x (10.22 + Hb concentration) / (1.7 x Hb concentration) Females: Hb corrected DLCO = measured DLCO x (9.38 + Hb concentration) / (1.7 x Hb concentration). Annual rate of decline in haemoglobin corrected diffusing capacity of the lung for carbon monoxide (DLCO) decrease is presented.
Time Frame: From first drug administration in 1199.35 until database lock 15Oct2015, up to 61.8 Months
Population: FAS
Measure: Mean (Standard Error); unit: mmol/min/kPa/yr
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
mmol/min/kPa/yr | -0.4 (0.08) | -0.3 (0.04) | -0.2 (0.07)

5. Secondary Outcome: Percentage of Patients With at Least One Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation
Description: Percentage of patients with at least one acute idiopathic pulmonary fibrosis (IPF) exacerbation are presented.
  An exacerbation was defined as otherwise unexplained clinical features occurring within
  1 month including all of the following:
  * Progression of dyspnoea over several days to 4 weeks
  * New diffuse pulmonary infiltrates on chest X-ray and/or high-resolution computerised tomography (HRCT) Parenchymal abnormalities with no pneumothorax or pleural effusion (new ground-glass opacities) since the last visit
  * A decrease in arterial oxygen partial pressure (PaO2) of ≥10 mmHg or PaO2/fraction of inspired oxygen (FiO2) of <225 mmHg since the last visit
  * Exclusion of infection based on routine clinical practice and microbiological studies
  * Absence of other contributory causes such as congestive heart failure, pulmonary embolism, etc.
Time Frame: From first drug administration in 1199.35 until database lock 15Oct2015, up to 61.8 Months
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
Percentage of participants | 13.5 (0.08) | 19.8 (0.04) | 20.0 (0.07)

6. Secondary Outcome: Incidence of Patients With at Least One Acute IPF Exacerbation Over Time
Description: Incidence rate = (Patients with at least one acute IPF exacerbation / Total number of years at risk) x 100
Time Frame: From first drug administration in 1199.35 until database lock 15Oct2015, up to 61.8 Months
Population: FAS
Measure: Number; unit: Exacerbations Per Year
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
Exacerbations Per Year | 6.1 (0.08) | 7.6 (0.04) | 7.8 (0.07)

7. Secondary Outcome: Time to First Acute IPF Exacerbation
Description: Due to rare events, the median of time to event is not calculable, thus Kaplan-Meier estimates (providing the percentage of patients without acute IPF exacerbation for a certain amount of time after treatment) and confidence intervals (using Greenwood variance formula) are reported and presented within each treatment arm as secondary endpoint.
Time Frame: From first drug administration in 1199.35 until database lock 15Oct2015, up to 61.8 Months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
percentage of participants | 67.7 (29.47) [39.4 to 95.9] | 68.6 (14.60) [56.8 to 80.4] | 73.5 (28.22) [55.9 to 91.1]

8. Secondary Outcome: Percentage of Patients With at Least One Adverse Events (AEs), With Investigator Defined Drug-Related AEs, AEs Leading to Discontinuation of Trial Drug, Serious AEs
Description: Percentage of patients with at least one Adverse events (AEs), with investigator defined drug-related AEs, AEs leading to discontinuation of trial drug, serious AEs are presented
Time Frame: From the first nintedanib intake in trial 1199.35 to the last nintedanib intake + 28 days; up to 61.8 months + 28 days
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Number analyzed (Participants) | 37 | 126 | 35
Percentage of participants
  AEs | 100.0 (0.08) | 99.2 (0.04) | 97.1 (0.07)
  Investigator defined drug-related AEs | 70.3 | 65.9 | 54.3
  AEs leading to discontinuation of trial drug | 48.6 | 41.3 | 34.3
  Serious AE | 67.6 | 74.6 | 62.9

ADVERSE EVENTS:
Time Frame: From the first nintedanib intake in trial 1199.35 to the last nintedanib intake + 28 days; up to 61.8 months + 28 days
Arm/Group | Placebo | Nintedanib 50 mg- 100 mg | Nintedanib 150 mg
Serious Adverse Events (participants affected / at risk) | 25/37 | 94/126 | 22/35
Other Adverse Events (participants affected / at risk) | 34/37 | 111/126 | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | Nintedanib 50 mg- 100 mg (N=126) | Nintedanib 150 mg (N=35)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 3 | 0
Angina unstable (Cardiac disorders) | 0 | 3 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Bundle branch block (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 5 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 1
Right ventricular failure (Cardiac disorders) | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 2 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 1
Death (General disorders) | 1 | 1 | 0
Disease progression (General disorders) | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Sudden death (General disorders) | 0 | 2 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 3 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 4 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 5 | 3
Pneumonia (Infections and infestations) | 3 | 6 | 2
Pneumonia escherichia (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 4 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pancreatic enzymes increased (Investigations) | 0 | 1 | 0
Troponin I (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Coma (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 11 | 41 | 10
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | Nintedanib 50 mg- 100 mg (N=126) | Nintedanib 150 mg (N=35)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0
Cataract (Eye disorders) | 2 | 9 | 3
Glaucoma (Eye disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 9 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 68 | 22
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4 | 2
Nausea (Gastrointestinal disorders) | 9 | 22 | 2
Vomiting (Gastrointestinal disorders) | 7 | 17 | 3
Chest pain (General disorders) | 2 | 10 | 1
Condition aggravated (General disorders) | 2 | 0 | 1
Fatigue (General disorders) | 2 | 9 | 4
Influenza like illness (General disorders) | 0 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2 | 2
Bronchitis (Infections and infestations) | 12 | 27 | 6
Cystitis (Infections and infestations) | 2 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 8 | 4
Influenza (Infections and infestations) | 1 | 9 | 6
Lower respiratory tract infection (Infections and infestations) | 4 | 12 | 1
Nasopharyngitis (Infections and infestations) | 8 | 24 | 6
Pneumonia (Infections and infestations) | 2 | 3 | 1
Respiratory tract infection (Infections and infestations) | 3 | 8 | 3
Sinusitis (Infections and infestations) | 0 | 9 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 2 | 2 | 0
Tracheobronchitis (Infections and infestations) | 2 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 10 | 1
Urinary tract infection (Infections and infestations) | 2 | 11 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 6 | 0
Hepatic enzyme increased (Investigations) | 2 | 3 | 0
Weight decreased (Investigations) | 10 | 29 | 7
Decreased appetite (Metabolism and nutrition disorders) | 6 | 17 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 10 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Dizziness (Nervous system disorders) | 4 | 11 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 4 | 3
Depression (Psychiatric disorders) | 2 | 4 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 3 | 2
Proteinuria (Renal and urinary disorders) | 1 | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 27 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 19 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 22 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Hypertension (Vascular disorders) | 0 | 7 | 3
Hypotension (Vascular disorders) | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.